CLINICAL TRIAL: NCT05979948
Title: A Prospective, Open-label, Multicenter Study of Zanubrutinib Combined With BR (Bendamustine/Rituximab) Regimen in Subjects With Newly-diagnosed Waldenström's Macroglobulinemia
Brief Title: A Phase 2 Clinical Trial to Evaluate Zanubrutinib Combined With BR (Bendamustine/Rituximab) Regimen in Subjects With Newly-diagnosed Waldenström's Macroglobulinemia
Acronym: CZ-WM01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: RenJi Hospital (Other); Huashan Hospital (Other); Shanghai 6th People's Hospital (Other); Huadong Hospital (Other)
Responsible Party: Principal Investigator, Juan Du, Director, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZ-WM01
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Waldenström's Macroglobulinemia
Keywords: Waldenström's macroglobulinemia; Zanubrutinib; BR regimen; newly-diagnosed
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanubrutinib combined with BR regimen (Experimental): Drug: zanubrutinib,160 mg oral capsules twice daily for 12 months Drug: Bendamustine,70-90 mg/m2 on days 1 and 2 of each cycle for 6 cycles. Drug: Rituximab,375 mg/m2 intravenously on day 0 of each cycle for 6 cycles.
  Interventions: Drug: Zanubrutinib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib, 160 mg oral capsules twice daily for 12 months
Drug: Bendamustine — Bendamustine, 70-90 mg/m2 on days 1 and 2 of each cycle for 6 cycles.
Drug: Rituximab — Rituximab, 375 mg/m2 intravenously on day 0 of each cycle for 6 cycles

SUMMARY:
This was a single-arm, multicenter, Phase 2 study to evaluate the efficacy of zanubrutinib combined with BR (Bendamustine/Rituximab) regimen in Chinese participants with newly-diagnosed Waldenström's macroglobulinemia who exhibited one or more of the criteria for requiring treatment based on consensus guidelines from the 11th International Workshop on Waldenström's Macroglobulinemia (IWWM). The investigators propose this combination will improve the deep remission compared to single Zanubrutinib or BR regimen and can be a time-limited regimen which will reduce the life-time therapy and benefit the patients.

DETAILED DESCRIPTION:
The study comprised an initial screening phase (up to 7 days), a single-arm treatment phase, and a follow-up phase. Subjects with newly-diagnosed Waldenström's macroglobulinemia can participate if all eligibility criteria are met. The participants will receive bendamustine and rituximab for 6 28-day cycles. Bendamustine will be given intravenously at 70-90 mg/m2 on days 1 and 2 of each cycle. Rituximab will be given on day 1 of each cycle (375 mg/m2 intravenously), Zanubrutinib will be given orally 160mg Bid per day, up to 12 months. The participants with WM will also have disease assessment with Lymph node ultrasound and abdominal ultrasound each cource, serum IgM, serum protein electrophoresis (SPE), immunofixation (IFA), and viscosity assessments will be measured serially. A bone marrow aspiration and biopsy flow cytometry examination will be done before treatment and at response assessment at cycle 6 and 12. Durability of response will also be assessed every 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

1. Newly diagnosed patients with waldenström's macroglobulinemia meeting at least one criterion for treatment according to consensus panel criteria from the eleventh IWWM.
2. ECOG score: 0-3 points, estimated survival time exceeding 3 months.
3. Did not receive any treatment for Waldenström's macroglobulinemia before screening, except for glucocorticoid therapy for autoimmune hemolysis.
4. No serious damage to main organs, and meet the following laboratory examination indicators: creatinine clearance rate≥40ml/min, total bilirubin≤1.5 times of the upper limit of normal range; AST and ALT≤2.5 times of the upper limit of normal range; Myocardial enzyme≤2 times of the upper limit of normal range; ECHO must demonstrate left ventricular ejection fraction (LVEF) within the normal range, and no ECG abnormality with clinical significance.
5. Neutrophil count≥1.5×10^9/L without growth factor therapy within 7 days before screening; Platelet count≥50×10^9/L without growth factor support or transfusion within 7 days before screening; Hemoglobin≥60 g/L without erythropoietin (EPO) support or transfusion within within 7 days before screening.
6. No history of paroxysmal atrial fibrillation or chronic persistent atrial fibrillation.
7. Able to swallow and Oral administration.
8. The subjects complete all screening and evaluations listed in all trial protocols.
9. The subjects who signed the informed consent form for chemotherapy.

Exclusion Criteria:

1. Waldenström's macroglobulinemia with amyloidosis or POEM syndrome
2. HIV positive, or patients with active hepatitis A, hepatitis B, and hepatitis C infection; Or the number of copies of hepatitis B virus>10^2.
3. Accompanied by other serious unstable diseases, including heart failure, renal failure, liver failure, hemorrhagic diseases, uncontrollable diabetes, etc.
4. In the past two years, the terminal organ was damaged due to autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or the systemic use of immunosuppressive or other systemic disease control drugs was required.
5. Serious infectious diseases (uncured pulmonary tuberculosis, pulmonary aspergillosis, etc.).
6. Other uncontrolled malignancies (excluding non Melanoma skin cancer, cervical cancer in situ, bladder cancer cancer and breast cancer with disease-free survival of more than 5 years).
7. Individuals with epilepsy, dementia, and other mental disorders who require medication treatment and are unable to understand or follow the research protocol.
8. Drug use, medical, psychological, or social conditions that may interfere with participants' participation in the study or evaluation of the results.
9. Pregnant and lactating women.
10. Patients who are accounted to be not appropriate for this trail by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of 12 cycles of treatment(each cycle is 28 days)
  ORR is defined as the percentage of participants with a minor, partial, very good partial, and complete response
The best deep response rate | Time Frame: up to the end of 12 cycles of treatment(each cycle is 28 days)
  defined as complete response (CR) and very good partial response (VGPR)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 6 years post first dose
  PFS was defined as from the initiation of treatmentuntil to first documentation of progression or death, whichever comes first.
Overall Survival (OS) | Up to 6 years post first dose
  OS is measured from the date of the initial of treatment to the date of the subject's death.
minimal residual disease (MRD) rate | Up to 6 years post first dose
  MRD will be assessed at two on treatment timepoints (before start of cycles 7, 12) and every 6 months thereafter. MRD will be measured through bone marrow samples using flow cytometrey.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Doctor, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No